CLINICAL TRIAL: NCT04151719
Title: An Open-Label Extension Study to Evaluate the Safety and Efficacy of Oral Methylnaltrexone Bromide Tablets in Subjects With Advanced Pancreatic Cancer
Brief Title: An Extension Study of Methylnaltrexone Bromide (MNTX) in Participants With Advanced Pancreatic Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to pandemic challenges and consideration of a different study design in the future.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAL-REL-2043
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MNTX 450 mg QD (Experimental): Participants will receive methylnaltrexone bromide (MNTX) 450 milligrams (mg) (3 tablets of 150 mg each) once daily (QD) orally. Treatment will continue until participant's death or early withdrawal from the study or study termination by the sponsor.
  Interventions: Drug: Methylnaltrexone bromide (MNTX)

INTERVENTIONS:
Drug: Methylnaltrexone bromide (MNTX) — Methylnaltrexone bromide will be administered per dose and schedule specified in the respective arm.
  Other Names: Relistor®

SUMMARY:
This open-label extension study will evaluate the long-term safety and efficacy of oral MNTX in participants with advanced pancreatic cancer (adenocarcinoma) who were previously enrolled in Study SAL-REL-2042 (NCT04083651).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants greater than or equal to (≥)18 years of age on the date the Informed Consent Form (ICF) is signed, with the capacity to provide voluntary informed consent.
* Enrolled in double-blind Study SAL-REL-2042 (NCT04083651) and completed an end of study (EOS) visit (Day 168) or completed Day 56 of the Study SAL-REL-2042 (NCT04083651).
* Must be able to read, understand, and provide written informed consent on the Institutional Review Board (IRB)-approved ICF and provide authorization, as appropriate, for local privacy regulations.
* Willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.
* Signed an informed consent/Health Insurance Portability and Accountability Act (HIPAA) form.

Exclusion Criteria:

* Concurrent therapy with any other investigational agent during the study.
* Current use of a peripherally acting mu-opioid-receptor antagonist.
* Current evidence of untreated brain metastasis(es).
* Diarrhea greater than Grade 1, based on the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0).
* Bowel obstruction.
* Advanced liver disease.
* Renal disease.
* Any other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Principal Investigator, would make the participant inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-03 (Estimated); Primary Completion 2024-02-03 (Estimated); Study Completion 2024-02-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From first MNTX dose administration until death from any cause (up to 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: John Lahey, Study Director — Bausch Health Americas, Inc.